CLINICAL TRIAL: NCT06250192
Title: A Randomized Controlled Trial Evaluating the Effect of Virtual Patient-centered Education on Infant Birthweight in Women With Diabetes Mellitus
Brief Title: Educational TOolS for Pregnant Women With Diabetes Mellitus
Acronym: ETOS-DM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2024-02-01; First posted 2024-02-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus; Pregnancy Complications
MeSH Terms: conditions — Diabetes Mellitus; Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with patient-centered virtuel educational tools (Experimental): Patient randomized to intervention with patient-centered virtuel educational tools based on small videos
  Interventions: Other: Virtuel education
- Control: Women were randomized to usal care (No Intervention): Randomized to standard treatment without acces to virutel educational tools

INTERVENTIONS:
Other: Virtuel education — Randomization to virtuel education based on a tool of small videos accessible via smartphones
  Arms: Intervention with patient-centered virtuel educational tools

SUMMARY:
A randomized controlled trial evaluating whether a patient-centered virtual educational tool based on small videos focusing on optimization of mental health, diet, physical activity, self-adjustment of insulin dose and use of diabetes technology in addition to usual individual face-to-face education, will improve glycemic control and pregnancy outcome in women with pre-existing diabetes mellitus compared to women receiving usual individual face-to-face education alone.

DETAILED DESCRIPTION:
ETOS-DM is a national RCT evaluating the effect of combined virtual patient-centered education based on a tool of small videos accessible via smartphones in addition to usual individual face-to-face education during pregnancy or to routine individual face-to-face education only.

The small educational videos covering topics as food choices, physical activity, self-adjustment of insulin dose insulin pump settings during pregnancy, use of CGM during pregnancy, mental health among others,each of 1-4 minutes duration, will be developed in collaboration with user representatives (women with pre-existing diabetes who are or have recently been pregnant) and relevant health care professionals.

The inclusion period of the ETOS-DM study starts on September 1st 2023 and ends on August 31st 2025.

Pregnant women with pre-existing diabetes will be randomized before 14 gestational weeks. The women in the intervention group will have free, unlimited access to approximately 10 educational videos. The use of these virtual educational videos will be monitored and the women's own experience with the videos will be explored. The women will be followed during pregnancy, delivery until one month after delivery. Both groups of women follow usual local care and local face-to-face education which is allowed to change during the study period.

Stratification will be performed for diabetes center, for diabetes type and, in women with type 1 diabetes, use of MDI or insulin pump.

ELIGIBILITY:
Inclusion Criteria:

* Women, age ≥ 18 years
* Type 1 diabetes, type 2 diabetes or other types of pre-existing diabetes (e.g., maturity onset diabetes of the young (MODY))
* Pregnant with one or more intrauterine singleton living foetus(es) (5 to 13 completed gestational weeks) at inclusion confirmed by an ultrasound scan)

Exclusion Criteria:

* A diagnosis with severe mental or psychiatric barriers or a concurrent disease based on the decision of the investigator
* No proficiency in Danish to understand oral and written information

To secure independent observations, women can be randomized in the ETOS-DM study only once.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Birthweight standard deviation score | At delivery
  Offspring birth weight adjusted for gestational age and gender (standard deviation (SD) score)

SECONDARY OUTCOMES:
HbA1c during pregnancy | At inclusion, at 21 weeks, at 33 weeks and at 35 weeks
  HbA1c levels during pregnancy at inclusion, 21, 33 and 35 weeks
Continuous glucose monitoring data | Throughout pregnancy and 1 month post delivery
  The average glucose level and percentage of time spent in the continuous glucose monitoring (CGM) target range 3.5-7.8 mmol/L, below target range (glucose <3.5 mmol/L) or above target range (glucose >7.8 mmol/L). The levels will be evaluated at night-time (24 pm to 6 am) and over 24 h, respectively, in pregnancy, during delivery and in the first one-month period after delivery.
  • The incidence of severe hypoglycemia in the year preceding pregnancy, during pregnancy and in the first one-month period after delivery
Severe hypoglycemia | 2 years
  The incidence of severe hypoglycemia in the year preceding pregnancy, during pregnancy and in the first one-month period after delivery
Maternal weight gain | At inclusion, at 21 weeks, at 33 weeks, 35 weeks and one month after delivery
  Maternal gestational weight gain and weight retention one month after delivery
Individuel insulin pump settings in women using insulin pump | At inclusion, at 21 weeks, at 33 weeks, 35 weeks, at delivery and one month after delivery
  In women using insulin pump the following will be collected: insulin pump settings at study visits, at delivery andthe first month after delivery during lactation
Fetal overgrowth | At birth
  The prevalence of fetal overgrowth, defined as the offspring birth weight SD score >90th percentile
Pregnancy complications | 9 months
  The prevalence of induced abortion (including indication for abortion), miscarriage, gestational hypertension, preeclampsia, need for maternal corticosteroid treatment for fetal lung maturation, diabetic ketoacidosis, urinary tract infection, early preterm delivery (before 34 completed weeks), preterm delivery (before 37 completed weeks), preterm prelabour rupture of the membranes
Prevalence of birth complications | At birth and one month post delivery
  The prevalence of shoulder dystocia, birth canal trauma, mode of delivery (vaginal, cesarean section, instrumental delivery), postpartum hemorrhage, maternal death, antihypertensive treatment given one month after delivery
Prevalence of neonatal morbidity | 1 month
  Neonatal morbidity (neonatal hypoglycemia, jaundice, respiratory distress, transient tachypnoea, duration of stay in neonatal intensive care unit, total number of admission days), cord blood pH, stillbirths, infant death within one month
Major congenital malformations | 9 months
  Number of major congenital malformations (ICD10 Q00-Q99 or requiring medical or surgical treatment)
Infant growth at one month of age | 1 month
  Infant growth and health at one month of age
Maternal reported outcomes during pregnancy and one month postpartum | In early pregnancy, in late pregnancy and one month post-partum.
  Maternal reported outcomes, including measures assessing health status (SF-12), depression (EPDS), well-being (WHO-5), pregnancy-specific worries (CWS), perceived stress (PSS), loneliness (T-ILS), diabetes related distress (PAID), fear of hypoglycaemia (HFS-II worry scale), satisfaction with care (PACIC), psychopathology developing during pregnancy and pre-natal attachment (MAAS).
Partner reported outcomes during pregnancy and one month postpartum | In early pregnancy, in late pregnancy and one month post-partum.
  Partner reported outcomes, including measures assessing health status (SF-12), depression (EPDS), well-being (WHO-5), pregnancy-specific worries (CWS), perceived stress (PSS), loneliness (T-ILS), diabetes related distress (PAID), fear of hypoglycaemia (HFS-II worry scale), satisfaction with care (PACIC), psychopathology developing during pregnancy and pre-natal attachment (MAAS).
Continuous glucose monitoring metrics 1 months post delivery | 1 months
  Average glucose level and the percentage of time in the first one-month period after delivery spent in the CGM target range 3.9-10.0 mmol/L, below target range (glucose <3.5 mmol/L) or above target range (glucose >7.8 mmol/L) at night-time (24 pm to 6 am) and over 24 h, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Mathiesen, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Center for Pregnant Women with Diabetes, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No